CLINICAL TRIAL: NCT05758181
Title: Undermining Apices in Surgical Wounds: a Randomized Evaluator-blinded Split-wound Comparative Effectiveness Trial
Brief Title: Undermining Apices in Surgical Wounds
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 1999193
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Scarring
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two blinded observers will record their scores independently using the POSAS instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linear Wound Closure (No Intervention): A cutaneous layer of sutures will be placed on one side, as is standard of care.
- Linear Wound Closure with Apical Undermining (Experimental): The other side of the wound will have a cutaneous layer of sutures, as is standard of care, and will receive apical undermining.
  Interventions: Other: Apical Undermining

INTERVENTIONS:
Other: Apical Undermining — The skin at the tip of the wound will be freed to reduce tension.
  Arms: Linear Wound Closure with Apical Undermining

SUMMARY:
When patients have surgery on the neck, trunk, arms, or legs, stitches are the standard way to close the wound. Wounds always result in a scar, but doctors are always looking for ways to reduce scarring. Several studies have been done to test ways to close wounds that reduce scarring. One idea is to reduce the tension around the cut. One way to reduce tension is to free up the skin around the wound. This procedure is also called "undermining". Some studies have shown that freeing up the skin near the tips of the wound, called the "apices," is helpful for improving the cosmetic outcome of scars. This study will investigate if there are any differences in the appearances of the scar if one tip is undermined and the other is not.

DETAILED DESCRIPTION:
Reducing scar tissue formation and postoperative complications in wound closure has remained the focus of recent studies and decreases the cost and time burden of follow-up visits and procedures. Such studies have highlighted the impact of mechanical forces and tension on scar formation, demonstrating that reducing the mechanical stress within the wound environment results in better aesthetic outcomes. Undermining peripheral and apices of the wound has been used in the closure of large and tight defects allowing the closure of these wounds by reducing the tension. Undermining has been shown to reduce tension, and peripheral and apical undermining has been recommended for decreasing scar formation. However, extensive undermining may increase the complications of the surgery by reducing vascularization and creating a space for hematomas. To our knowledge, the impact of scar cosmesis and the rate of postoperative complications in apical undermining in the linear repair of surgical wounds have not been studied, and it remains unknown whether undermining the apices can decrease the protrusion of the scar tissue at the edges. This study seeks to determine the effectiveness of apical undermining of linear wound closures in improving scar cosmesis by using individuals as their own controls in a split-scar model.

This is a single center, randomized, evaluator-blinded, split wound study.

After screening and informed consent, demographic data will be collected including age, race, gender, and medical record number. This will be collected within the Redcap database.

The patient's wound will be labeled A if it is on the left or superior side of the investigator and B if it is on the right or inferior side. A concealed randomization result will be obtained from the Redcap randomization module, which will specify which side, A or B, will receive apical undermining

Following this, both sides of the wound will be sutured together with a subcutaneous (bottom) layer of stitches. Next, a cutaneous layer of sutures will be placed, as is the standard of care. A digital image of the wound after the epidermal closure will be obtained; these may be used in scientific talks and/or for publication purposes. The patient will then be instructed to continue dressing changes along the entire length of the surgical site until the wound is fully healed as is the standard of care.

Treatment assignment, wound length, demographic data, and digital images will be recorded within the Redcap database. Follow-up assessment will be scheduled for three months following the procedure, with a one-month window before or after that time if the patient cannot return at precisely three months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the neck, trunk, and extremities with predicted primary closure
* Willing to return for follow-up visit

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant women
* Unable to understand written and oral English
* Wounds with predicted closure length less than 3cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Observer Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  The primary endpoint will be the score of two blinded reviewers independently using the POSAS assessment. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability, and surface area). All items are scored on a scale ranging from 1 ("like normal skin") to 10 ("worst scar imaginable"). The sum of the six items results in a total score of the POSAS observer scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.

SECONDARY OUTCOMES:
Patient Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  This is the patient portion of the POSAS assessment, which will be independently recorded. The patient scale of the POSAS consists of six items (pain, itch, thickness, color, stiffness, and irregularity). All items are scored on a scale ranging from 1 ("as normal skin") to 10 ("yes, very different"). The sum of the six items results in a total score of the POSAS patient scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10.
Width of Scar as measured using Trace-to-Tape Method | 3 months
  The trace-to-tape method is an objective measure for linear postoperative scars. The mean scar width will be determined using the trace-to-tape method. The surface area of the scar will be collected by tracing the scar with a water-based gel pen. While still wet, the gel residue will be lifted from the skin with clear packing tape and transferred on a sheet of paper.
Complications or Adverse Events from Treatment | 3 months
  For example, if one half of the scar has more associated erythema, as measured using the Trace-to-Tape method, then it will be recorded. Other complications from the treatment will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis - Dermatology
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States

REFERENCES:
- [Background] Gurtner GC, Dauskardt RH, Wong VW, Bhatt KA, Wu K, Vial IN, Padois K, Korman JM, Longaker MT. Improving cutaneous scar formation by controlling the mechanical environment: large animal and phase I studies. Ann Surg. 2011 Aug;254(2):217-25. doi: 10.1097/SLA.0b013e318220b159. PMID 21606834
- [Background] Barnes LA, Marshall CD, Leavitt T, Hu MS, Moore AL, Gonzalez JG, Longaker MT, Gurtner GC. Mechanical Forces in Cutaneous Wound Healing: Emerging Therapies to Minimize Scar Formation. Adv Wound Care (New Rochelle). 2018 Feb 1;7(2):47-56. doi: 10.1089/wound.2016.0709. PMID 29392093
- [Background] Krishnan NM, Brown BJ, Davison SP, Mauskar N, Mino M, Jordan MH, Shupp JW. Reducing Wound Tension with Undermining or Imbrication-Do They Work? Plast Reconstr Surg Glob Open. 2016 Jul 13;4(7):e799. doi: 10.1097/GOX.0000000000000799. eCollection 2016 Jul. PMID 27536478
- [Background] Zitelli JA. TIPS for a better ellipse. J Am Acad Dermatol. 1990 Jan;22(1):101-3. doi: 10.1016/0190-9622(90)70016-b. PMID 2405023
- [Background] Jonathan K (Ed). Dermatologic Surgery. McGraw-Hill Education. 2018. ISBN: 978-1-25-964392-7.